CLINICAL TRIAL: NCT03207477
Title: Visual Maturation in Prematurely Born Infants According to Factors Influencing Its Development. Premavision Follow-up at 18 Months Corrected Age, 4 and 7 Years of Age.
Brief Title: Premavision Cohort Follow-up
Acronym: PrmvsionSuiv
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator not available anymore (Sabbatical)
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016-A02017-44
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Visual Disorder
Keywords: Infant; Prematurely born; maturation
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: Longitudinal cohort study with a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prematurely born infants (Experimental): Visual acuity measurement in prematurely born infants included in PREMAVISION study
  Interventions: Diagnostic Test: Visual acuity measurement
- Term born infants (Active Comparator): Visual acuity measurement in term born control infants
  Interventions: Diagnostic Test: Visual acuity measurement

INTERVENTIONS:
Diagnostic Test: Visual acuity measurement — visual acuity measurement by Baby Vision cards at 18 months corrected age, by Rossano Weiss test at 4 years of age and optometric tests of Parinaud and Snellen at 7 years of age
  Other Names: Measurement of cycloplegic refraction

SUMMARY:
This study aim at following a cohort of prematurely born infants at 18 months corrected age, 4 and 7 years of age. This cohort had an evaluation of visual maturation at term equivalent age (TEA) with factors associated with impaired visual maturation. (PREMAVISION-CLinicalTrials.gov ID: NCT02890251).

In this follow-up study, prematurely born infants vision will be compared to term born infants matched for postnatal age.

ELIGIBILITY:
Inclusion Criteria:

* Infants included in the Premavision cohort
* Term born healthy control infants at matched postnatal age

Exclusion Criteria:

* Ocular malformation
* Genetic abnormality
* Neurodevelopmental impairment

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity measurement | 18 months corrected age
  Baby Vision Cards
Visual acuity measurement | 4 years post-natal age
  Rossano Weiss test
Visual acuity measurement | 7 years post-natal age
  Parinaud and Snellen tests

SECONDARY OUTCOMES:
Measurement of cyclopegic refraction | 18 months corrected age
  Non invasive refraction measurement by autorefractometer Cycloplégie par Skiacol
Measurement of cyclopegic refraction | 4 years of age
  Non invasive refraction measurement by autorefractometer
Measurement of cyclopegic refraction | 7 years of age
  Non invasive refraction measurement by autorefractometer

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: No